CLINICAL TRIAL: NCT03458767
Title: A Cognitive Self-Management Intervention for Persons With Multiple Sclerosis: Adapting Web-based Technology
Acronym: PALMS-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2017-08-0062
Record Dates: First submitted 2017-11-21; First posted 2018-03-08 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Multiple Sclerosis
Keywords: Cognitive function; Physical activity; Self-management
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity

STUDY DESIGN:
Intervention Model Description: This pilot feasibility study employs a mixed methods design conducted in a community setting. Phase 1 uses a single-group qualitative design involving a convenience sample of 5 adults with MS; Phase 2 uses a randomized controlled trial (RCT) design conducted with a sample of 20 adults with MS (10 intervention/10 control). Phase 2 data will be collected at baseline (before the intervention) and at 8-weeks (post-intervention). Data includes self-report measures, an objective measure of physical activity, and neurocognitive tests. An "enhanced usual care" control group is selected as most appropriate for this pilot feasibility study of a non-pharmacologic, behavioral intervention.
Who Masked: Outcomes Assessor
Masking Description: A trained research assistant, blinded to the participant's group assignment, will collect the NIH Toolbox measures using an iPad at baseline and 8-weeks (post-intervention).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Eight weekly 90-minute group educational sessions attended via a computer, tablet, or smart phone using a web-based video conference platform.
  Interventions: Behavioral: Eight weekly 90-minute group educational sessions
- Control group (No Intervention): Enhanced usual care control group will receive an illustrated instructional booklet on Physical Activity for persons with MS developed by the National Center on Health, Physical Activity and Disability (NCHPAD).

INTERVENTIONS:
Behavioral: Eight weekly 90-minute group educational sessions — Eight weekly 90-minute group educational sessions, originally developed for the MAPSS-MS intervention, adapted for remote web-based delivery.
  Arms: Intervention group

SUMMARY:
Development and pilot testing of a cognitive self-management intervention for persons with multiple sclerosis (PwMS) emphasizing physical activity (PA) delivered via web-based video conference.

DETAILED DESCRIPTION:
The primary objective of this study is to develop and pilot test an innovative cognitive self-management intervention for PwMS delivered via web-based video conferencing. Data derived from interviews will be used to guide the adaptation of Stuifbergen's 8-week Memory, Attention, and Problem-Solving Skills in MS (MAPSS-MS) intervention to be delivered via web-based video conferencing. The adapted MAPSS-MS intervention will be feasibility tested in small groups of PwMS. Outcome variables include: (1) neurocognitive function assessed using the NIH Toolbox®, a comprehensive set of psychometrically sound neuro-behavioral measures that quickly assesses cognitive functions using an iPad, (2) objective PA and sleep using Actigraph™ accelerometers, (3) self-reported sleep, depression, and fatigue using the Patient-Reported Outcome Measurement Information System (PROMIS), and (4) MS specific self-management using the Multiple Sclerosis Self-Management Scale (MSSM). Community-residing PwMS, age 21 to 70, will be recruited from Central Texas to participate in Phase 1 interviews (n=5) and Phase 2 pilot testing (n=20) of the adapted version of the 8-week MAPSS-MS cognitive self-management intervention emphasizing PA delivered via web-based video conferencing. In Phase 2 pilot testing (n=20), an intervention group (n=10) will be compared to an "enhanced usual care" control group (n=10).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of clinically definite MS documented by their healthcare provider
* Age 21 to 70
* Capable of understanding and complying with the study protocol
* Able to read and write in English
* Stable disease at the time of entry into the study (relapse free for at least 90 days)
* Willing to participate in an 8-week study promoting physical activity, MS self-management and compensatory cognitive strategies, and data collection
* Have subjective concerns about their cognitive functioning (score ≥ 10 on the 20-item Perceived Deficits Questionnaire)
* Any gender
* Any ethnic/racial group

Exclusion Criteria:

* Currently pregnant or plan to be
* Diagnosed with cardiovascular or respiratory disease, other medical causes of dementia or other neurological disorders that may impact cognition or emotions
* Evidence of major psychiatric disorder
* Major functional limitations that preclude them from participating in the study

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline NIH Toolbox Picture Vocabulary Test at 8-weeks (post-intervention) | Baseline and 8-weeks (post intervention)
  Test of vocabulary knowledge
Change from Baseline NIH Toolbox Oral Reading Recognition at 8-weeks (post-intervention) | Baseline and 8-weeks (post intervention)
  Test of oral reading (decoding) skills
Change from Baseline NIH Toolbox Flanker Inhibitory Control and Attention Test at 8-weeks (post-intervention) | Baseline and 8-weeks (post intervention)
  Test of executive function - the capacity to plan, organize and monitor the execution of behaviors that are strategically directed in a goal-oriented manner) and attention (allocation of one's limited capacities to deal with an abundance of environmental stimulation) test.
Change from Baseline NIH Toolbox Dimensional Change Card Sort Test at 8-weeks (post-intervention) | Baseline and 8-weeks (post intervention)
  Test of attention - the allocation of one's limited capacities to deal with an abundance of environmental stimulation) test.
Change from Baseline NIH Toolbox List Sorting Working Memory Test at 8-weeks (post-intervention) | Baseline and 8-weeks (post intervention)
  Test of working memory - the capacity of an individual to hold information in a short-term buffer and manipulate the information.
Change from Baseline NIH Toolbox Oral Symbol Digit Test at 8-weeks (post-intervention) | Baseline and 8-weeks (post intervention)
  Test of processing speed - the amount of time it takes to mentally process a set amount of information, or the amount of information that can be processed within a certain unit of time. It is a measure that reflects mental efficiency.
Change from Baseline NIH Toolbox Pattern Comparison Processing Speed Test at 8-weeks (post-intervention) | Baseline and 8-weeks (post intervention)
  Test of processing speed - the amount of time it takes to mentally process a set amount of information, or the amount of information that can be processed within a certain unit of time. It is a measure that reflects mental efficiency.
Change from Baseline NIH Toolbox Picture Sequence Memory Test at 8-weeks (post-intervention) | Baseline and 8-weeks (post intervention)
  Test of episodic memory - the acquisition, storage and retrieval of new information. It involves conscious recollection of information learned within a context.

SECONDARY OUTCOMES:
Change from Baseline Multiple Sclerosis Self-Management Scale (MSSM) at 8-weeks (post-intervention) | Baseline and 8-weeks (post intervention)
  A 24-item self-report instrument developed specifically to address self-management in persons with MS.
Change from Baseline PROMIS Short Form v1.0 - Self-Efficacy for Managing Medications and Treatments 4a at 8-weeks (post-intervention) | Baseline and 8-weeks (post intervention)
  A 4-item self-report measure of confidence in managing medication schedules of different complexity. Items also assess managing medication and other treatments in challenging situations such as when traveling, when running out of medication, and when adverse effects are encountered.
Change from Baseline PROMIS Short Form v1.0 - Self-Efficacy for Managing Symptoms 4a at 8-weeks (post-intervention) | Baseline and 8-weeks (post intervention)
  A 4-item self-report measure of confidence to manage/control symptoms, to manage symptoms in different settings (home, public place, an unfamiliar place) and to keep symptoms from interfering with work, sleep, relationships or recreational activities.
Change from Baseline PROMIS Short Form v1.0 - Self-Efficacy for Managing Daily Activities 4a at 8-weeks (post-intervention) | Baseline and 8-weeks (post intervention)
  A 4-item self-report measure of confidence in performing various activities of daily living (ADLs) without assistance. Items also assess exercise, sexual activities and managing activities in challenging situations (traveling, bad weather).
Change from Baseline Neuro-Quality of Life (QoL) Short Form v2.0 - Cognitive Function at 8-weeks (post-intervention) | Baseline and 8-weeks (post intervention)
  An 8-item self-report measure of mental acuity, concentration, verbal and nonverbal memory, verbal fluency, and perceived changes in these cognitive functions.
Change from Baseline Neuro-QoL Short Form v1.0 - Depression at 8-weeks (post-intervention) | Baseline and 8-weeks (post intervention)
  An 8-item self-report measure of negative mood (sadness, guilt), views of self (self-criticism, worthlessness), and social cognition (loneliness, interpersonal alienation), as well as decreased positive affect and engagement (loss of interest, meaning, and purpose). Somatic symptoms (changes in appetite, sleeping patterns) are not included, which eliminates consideration of these items' confounding effects when assessing patients with comorbid physical conditions. Assesses depression over the past seven days.
Change from Baseline Neuro-QoL Short Form v1.0 - Fatigue at 8-weeks (post-intervention) | Baseline and 8-weeks (post intervention)
  An 8-item self-report measure of fatigue symptoms, from mild subjective feelings of tiredness to an overwhelming, debilitating, and sustained sense of exhaustion that likely decreases one's ability to execute daily activities and function normally in family or social roles. Fatigue is divided into the experience of fatigue (frequency, duration, and intensity) and the impact of fatigue on physical, mental, and social activities. Assesses fatigue over the past seven days.
Change from Baseline Neuro-QoL Short Form v1.0 - Sleep Disturbance 4a at 8-weeks (post-intervention) | Baseline and 8-weeks (post intervention)
  An 8-item self-report measure of sleep quality, sleep depth, and restoration associated with sleep. This includes perceived difficulties and concerns with getting to sleep or staying asleep, as well as perceptions of the adequacy of and satisfaction with sleep. Sleep Disturbance does not focus on symptoms of specific sleep disorders, nor does it provide subjective estimates of sleep quantities (total amount of sleep, time to fall asleep, amount of wakefulness during sleep). Assesses sleep disturbance over the past seven days.
Change from Baseline Physical Activity - steps at 8-weeks (post-intervention) | Baseline and 8-weeks (post intervention)
  Accelerometer step count
Change from Baseline Physical Activity - activity count at 8-weeks (post-intervention) | Baseline and 8-weeks (post intervention)
  Accelerometer activity count
Change from Baseline Sleep quality - sleep latency at 8-weeks (post-intervention) | Baseline and 8-weeks (post intervention)
  Accelerometer sleep latency
Change from Baseline Sleep quality - wake after sleep onset at 8-weeks (post-intervention) | Baseline and 8-weeks (post intervention)
  Accelerometer wake after sleep onset
Change from Baseline Sleep quality - total sleep time at 8-weeks (post-intervention) | Baseline and 8-weeks (post intervention)
  Accelerometer total sleep time
Change from Baseline Sleep quality - sleep efficiency at 8-weeks (post-intervention) | Baseline and 8-weeks (post intervention)
  Accelerometer sleep efficiency

CONTACTS AND LOCATIONS:
Overall Officials: Janet D Morrison, PhD, Principal Investigator — The University of Texas at Austin
Locations (1):
- The University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data from this pilot study

DOCUMENTS (2):
  • Study Protocol (2017-09-19): https://cdn.clinicaltrials.gov/large-docs/67/NCT03458767/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-19): https://cdn.clinicaltrials.gov/large-docs/67/NCT03458767/SAP_001.pdf